CLINICAL TRIAL: NCT01688661
Title: The Effects of Age and Gender on the Advantage of Sniffing Position for Laryngoscopic View
Status: Completed | Type: Observational
Sponsor: Kyung Hee University Hospital at Gangdong (Other)
Responsible Party: Principal Investigator, Jong-Man Kang, Associate professor, Kyung Hee University Hospital at Gangdong
Other Study IDs: KHNMC 2012-074
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Laryngeal View

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

SUMMARY:
The sniffing position has been regarded as a standard position for direct laryngoscopic view. This study evaluated the effects of the age and gender on the advantage of the sniffing position compared with simple head extension for laryngeal view during direct laryngoscopy.

ELIGIBILITY:
Inclusion Criteria:

* • Patients who are scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* • Patients with anatomical defects of the face, neck, or upper airway

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients who are scheduled for elective surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
the percentage of glottic opening | during laryngoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Kyung Hee University Gangdong Hospital, Seoul, South Korea